CLINICAL TRIAL: NCT02680834
Title: Randomized Trial Comparing a Dual Action Pneumatic Compression System Against Multi-Layer Bandaging Systems: A Non-Inferiority Study
Brief Title: VLU Non-Inferiority Study Comparing a Dual Action Pneumatic Compression Device to Multi-Layer Bandaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The ACT was re-designed per physician feedback and patient compliance & not because of safety.
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6010
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-01

CONDITIONS: Venous Leg Ulcer
Keywords: venous stasis ulcer; wound; chronic venous insufficiency
MeSH Terms: conditions — Varicose Ulcer; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual Action Pneumatic Compression Device (Experimental): ACTitouch dual action pneumatic compression system used daily during wakeful hours for up to 16 weeks.
  Interventions: Device: Dual Action Pneumatic Compression Device
- Multi-layer bandaging (Active Comparator): PROFORE or Coban 2 to be worn 24 hours daily for up to 16 weeks.
  Interventions: Device: Multi-Layer Bandaging

INTERVENTIONS:
Device: Dual Action Pneumatic Compression Device — Dual action pneumatic compression device used to treat chronic VLUs.
  Other Names: ACTitouch system
  Arms: Dual Action Pneumatic Compression Device
Device: Multi-Layer Bandaging — Multi-layer bandaging used to treated chronic VLUs
  Other Names: Profore or Coban 2
  Arms: Multi-layer bandaging

SUMMARY:
The purpose of the study is to test non-inferiority of chronic Venous Leg Ulcer (VLU) area reduction at 16 weeks with a dual action pneumatic compression device compared to multi-layer bandaging.

DETAILED DESCRIPTION:
Participants with a chronic venous leg ulcer will participate in a 2 week run in phase using standard of care multi-layer bandaging before being randomly assigned to either treatment using a dual action pneumatic compression device or continued multi-layer bandaging for up to 16 weeks. Participants will be seen in clinic for treatment and evaluation of symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years of age or legal age at the time of enrollment.
* Chronic venous insufficiency confirmed by ultrasound within previous 12 months or prior to randomization: if subject had bilateral CVI, the limb that possessed the largest ulcer meeting study criteria was used as the study treatment limb for evaluation and documentation throughout the study. Non-study limbs received standard of care treatment as determined by the treating clinician.
* Must have at least one of the following within the past six (6) months: Dorsalis Pedis (DP) systolic pressure ≥ 80mmHg for diabetic patients or ≥ 60mmHg for non-diabetic patients on study limb; Posterior Tibial (PT) systolic pressure ≥ 80mmHg for diabetic patients or ≥ 60mmHg for non-diabetic patients on study limb; Transcutaneous partial pressure oxygen (TcP02) > 30mmHg; Great toe systolic pressure > 40mmHg.
* Active ulceration (CEAP classification of C6): VLU was defined by open skin lesion of the leg or foot that occurred in an area affected by venous hypertension.
* Ulcer duration: Non healing VLU ≥ 1 month but not greater than 24 months.
* Ulcer size ≥ 2cm² ≤ 50cm²: if there were multiple ulcers on the study limb, the largest ulcer was used as the study treatment ulcer for evaluation and documentation throughout the study. If two ulcers were separated by no more than one centimeter of normal skin, their areas were added together for study purposes.
* Three or fewer separate full thickness ulcers on the study limb: sum of the ulcer areas on the study limb must be ≤ 50 cm².
* Leg circumferences within the following range: Ankle - 12 to 44cm; Calf - 22 to 60cm; Below knee - 22 to 68cm.
* Able and willing to provide informed consent prior to study participation.

Exclusion Criteria:

* Target ulcer or any other ulcer on the study limb involves exposure of tendon, muscle, or bone.
* Target ulcer was of non-venous etiology (sickle cell anemia, necrobiosis lipoidica diabeticorum, pyoderma, malignancy).
* Treatment of the target ulcer with living cellular therapy within 30 days of the time of projected randomization.
* Endovenous ablation or other venous surgery within two weeks of enrollment: venous ultrasound must be completed after procedure to determine whether there is still venous insufficiency at the time of enrollment.
* History of skin sensitivity to any of the components of ACT, multi-layer bandages of compression garments.
* History of an acute deep vein thrombosis (DVT) or pulmonary embolism (PE) within the last three (3) months.
* Acute thrombophlebitis within the last six (6) weeks.
* History of pulmonary edema or decompensated congestive heart failure within six (6) weeks of screening.
* Currently has an active infection of the skin on the target limb such as cellulitis requiring antibiotics.
* History of target limb cancer within the last 2 years with the exception of treated non-melanoma skin cancer unless ulcer biopsy performed at screening is negative for neoplasia.
* Active cancer receiving chemotherapy and/or radiation therapy.
* Poorly controlled diabetes with an HbA1c value of > 12% within the past three (3) months.
* Changes to medications that affected edema within the last 30 days prior to enrollment (e.g., diuretics, calcium channel blockers of the dihyropyridine class, pioglitazone, cox-1 inhibitors, pregabalin, and gabapentin, diltiazem, or fluctuating doses of systemic steroids).
* Use of systemic corticosteroids requiring daily administration at doses greater than 5mg of Prednisone per day or equivalent for greater than 2 weeks: low dose steroid administration (Prednisone up to 5 mg per day or equivalent) was allowable for an unlimited period of time. Topical steroid administration to peri-ulcer area or other skin was allowable but could not be applied to the ulcer itself.
* Currently pregnant or trying to become pregnant.
* Inability or unwillingness to participate in all aspects of study protocol.
* Exhibited any condition which, according to the Investigator, justified the subject's exclusion from the study, such as a medical condition where an increase in venous or lymphatic return is undesirable.
* Currently participating in another clinical trial.

Additional Exclusion Criteria after two week run-in:

* Subject's target ulcer decreased in size by greater than 30% compared to the baseline area.
* Subject's target ulcer increased in size by greater than 50% compared to the baseline area.
* Subject's target ulcer measured less than 1.5cm² at the Randomization Visit.
* Subject appeared to have evidence of infection in any ulcer.
* The sum of the ulcer areas on the subject's study limb is > 50cm².

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Marston, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (18):
- United States (18):
  - Phoenix VA Health Care System, Phoenix, Arizona
  - Associated Foot and Ankle Specialists, LLC, Phoenix, Arizona
  - Arizona Regional Medical Research, Tucson, Arizona
  - ILD Research Center, Carlsbad, California
  - Limb Preservation Platform - Northwest, Fresno, California
  - Limb Preservation Platform - Downtown, Fresno, California
  - Long Beach VA Healthcare System, Long Beach, California
  - UCLA Medical Center, Los Angeles, California
  - Greater Los Angeles VA Healthcare System, Los Angeles, California
  - VA San Diego Healthcare System, San Diego, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - University of Miami, Miami, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - Foot and Ankle Institute of South Florida, South Miami, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Stony Brook University, Stony Brook, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Jobst Vascular Institute, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marston WA, Kirsner RS, Tallis A, Hanft JR, Walters J, Farber A; ACTitouch Investigators. Economic benefit of a novel dual-mode ambulatory compression device for treatment of chronic venous leg ulcers in a randomized clinical trial. J Vasc Surg Venous Lymphat Disord. 2020 Nov;8(6):1031-1040.e1. doi: 10.1016/j.jvsv.2020.03.004. Epub 2020 May 22. PMID 32451241

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects participated in a two week run-in phase. The treatment included MLB which was worn 24 hours a day except during clinic visits. The run-in phase was intended to assess the subject's initial response to standard of care treatment using MLB before receiving treatment with the investigational device.
Period: Overall Study
Arm/Group | Dual Action Pneumatic Compression Device | Multi-layer Bandaging
Started | 26 | 30
Completed | 15 | 27
Not Completed | 11 | 3
Not completed — Physician Decision | 5 | 2
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dual Action Pneumatic Compression Device | Multi-layer Bandaging | Total
Number analyzed (Participants) | 26 | 30 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10) | 64 (10) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 17 | 23 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 17 | 23 | 40
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 21 | 23 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of VLU Area Reduction
Description: Percentage of ulcer area reduction in the target VLU during the 16 week treatment period calculated by wound imaging software.
Time Frame: Changes from Baseline to 16 weeks
Population: *Per Protocol Population (MITT patients who were randomized, received treatment, and did not exit the study early).
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Dual Action Pneumatic Compression Device | Multi-layer Bandaging
Number analyzed (Participants) | 13 | 24
percentage change | -83.8 (27.8) | -70.5 (52.0)

2. Secondary Outcome: Patient-Reported Quality of Life
Description: The Charing Cross Venous Ulcer Questionnaire assesses the patients' perception of their health when venous ulceration is present. All items are scored so that a lower score defines a more favorable health state (a greater reduction is associated with improved quality of life). In addition, each item is scored using a 1 to 5 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: Changes from Baseline to 16 weeks
Population: Per Protocol Population (Patients randomized who received treatment and had both Baseline and end of study measures).
Measure: Mean (Standard Deviation); unit: Change in total score
Arm/Group | Dual Action Pneumatic Compression Device | Multi-layer Bandaging
Number analyzed (Participants) | 15 | 27
Change in total score | -10.3 (15.4) | -1.7 (11.2)

3. Secondary Outcome: Outpatient Costs
Description: Assessment of the effect of the Actitouch compared to a standard regimen of multi-layer bandaging on mean total outpatient costs per subject.
Time Frame: Changes from Baseline to 16 weeks
Population: Per Protocol Population (Patients randomized who received treatment and had baseline and end of study measures).
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Dual Action Pneumatic Compression Device | Multi-layer Bandaging
Number analyzed (Participants) | 15 | 27
Dollars | 6748 (1308) | 8925 (2176)

ADVERSE EVENTS:
Time Frame: 16 Weeks
Description: An adverse event (AEs) includes any complication whose clinical significance is greater than anticipated, or which occurs with a frequency greater than that which is usually seen for this type of device.
Arm/Group | Dual Action Pneumatic Compression Device | Multi-layer Bandaging
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/26 | 2/30
Other Adverse Events (participants affected / at risk) | 17/26 | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Action Pneumatic Compression Device (N=26) | Multi-layer Bandaging (N=30)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lumbar stenosis; spondylolisthesis (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dual Action Pneumatic Compression Device (N=26) | Multi-layer Bandaging (N=30)
Pain/Discomfort (Nervous system disorders) | 3 | 6
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Infection (Infections and infestations) | 3 | 4
Ulcer (Skin and subcutaneous tissue disorders) | 4 | 5
Blister (Skin and subcutaneous tissue disorders) | 2 | 0
Other (General disorders) | 7 | 3

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects analyzed. Study was terminated early so the device could undergo a complete re-design to address physician feedback collected during the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multi-center publication, or if no multi-center publication is submitted for publication within 12 months after the conclusion or termination of the study at all sites, site may publish on your own site's data only. A draft of the manuscript must be submitted to Sponsor for review at least 45 days prior to submission for publication and 15 days for oral presentation. Sponsor shall respond to institution within 45 days of the receipt of draft.

DOCUMENTS (2):
  • Study Protocol (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT02680834/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT02680834/SAP_001.pdf